CLINICAL TRIAL: NCT01630694
Title: Three -Dimensional (3-D) Craniofacial Phenotyping of Patients With Difficult Airway
Brief Title: Three-dimensional Craniofacial Phenotyping of Patients With Difficult Airway
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study stopped due to not meeting enrollment goal.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jacek Wojtczak, Principal investigator, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RSRB case number: 00032136
Record Dates: First submitted 2011-08-16; First posted 2012-06-28 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Failed or Difficult Intubation
Keywords: Difficult airway management; anesthesia; difficult intubation
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Difficult intubation patients (Active Comparator): patients who were difficult to intubate during previous anesthetics provided by the staff anesthesiologists.
  Interventions: Procedure: 3D Laser Scanning of the Head; Procedure: Measurements and Digital Photo's of the head, neck and Mouth; Procedure: Ultrasound Exam of the Tongue
- Control (Placebo Comparator): The control group will consist of patients with the easy laryngoscopy and intubation, recruited prospectively.
  Interventions: Procedure: 3D Laser Scanning of the Head; Procedure: Measurements and Digital Photo's of the head, neck and Mouth; Procedure: Ultrasound Exam of the Tongue

INTERVENTIONS:
Procedure: 3D Laser Scanning of the Head — Five scans will be collected from different angles, each scan taking approximately 3 seconds. Each scan will consist of a thin beam of light flashing of your head.
  Other Names: Konica Minolta 3D Digitizing Konica Minolta 3D laser scanner
  Arms: Control
Procedure: Measurements and Digital Photo's of the head, neck and Mouth — Prior to the photographs, certain bone and soft tissue areas such as angle of the jaw, neck and chin will be gently touched and marked with self-adhesive paper stickers. Using the self-adhesive paper stickers and a measuring tape, we obtain measurements of your head and neck. You will be also asked to open your mouth and a digital photograph of the back of the mouth will be taken, as well as, pictures of the front and side of the head and neck.
  Other Names: General Electric Total access ultrasound
  Arms: Control
Procedure: Ultrasound Exam of the Tongue — The ultrasound study of the tongue will be performed after the series of laser scans. You will be examined in the sitting position. A small,handheld, curved ultrasound instrument will be placed under the chin to take images of the tongue. This exam should take less than a minute
  Other Names: General Electric Total access ultrasound
  Arms: Control
Procedure: 3D Laser Scanning of the Head — Five scans will be collected from different angles, each scan taking approximately 3 seconds. Each scan will consist of a thin beam of light flashing of your head.
  Other Names: 3D digitizing Konica Minolta 3D laser scanner
  Arms: Difficult intubation patients
Procedure: Measurements and Digital Photo's of the head, neck and Mouth — Prior to the photographs, certain bone and soft tissue areas such as angle of the jaw, neck and chin will be gently touched and marked with self-adhesive paper stickers. Using the self-adhesive paper stickers and a measuring tape, we obtain measurements of your head and neck.Digital Photographs of your Mouth - You will be also asked to open your mouth and a digital photograph of the back of the mouth will be taken, as well as, pictures of the front and side of the head and neck.
  Other Names: 3D digitizing konica minolta 3D laser scanner
  Arms: Difficult intubation patients
Procedure: Ultrasound Exam of the Tongue — The ultrasound study of the tongue will be performed after the series of laser scans. You will be examined in the sitting position. A small,handheld, curved ultrasound instrument will be placed under the chin to take images of the tongue. This exam should take less than a minute.
  Other Names: General Electric Total Access ultrasound
  Arms: Difficult intubation patients

SUMMARY:
The purpose of this study is to identify differences in craniofacial morphology and tongue size between patients who have a history of difficult airway management and a control group of patients who had an uneventful airway management during induction of general anesthesia. In this study the investigators want to validate the hypothesis that there are craniofacial phenotypic differences between patients who have a history of difficult airway management and a control group of patients who have had an uneventful airway management during the induction of general anesthesia.

DETAILED DESCRIPTION:
Difficult airway management is one of the most challenging tasks for anesthesiologists. Recent data from the American Society of Anesthesiologists (ASA) Management Closed Claims Project [1] show that the percentage of claims resulting from adverse respiratory events, though on the decline (42% in the 1980s to 32% in the 1990s), continue to constitute a large source of morbidity and mortality in anesthetized patients. In 2005, a closed claims analysis of trends in anesthesia-related death and brain damage between 1975 and 2000 showed that out of all respiratory events (n=503) responsible for death and brain damage, difficult endotracheal intubation (n=115), inadequate oxygenation (n=111) and inadvertent esophageal intubation (n=66) were the top three causes [2].

ELIGIBILITY:
Inclusion Criteria:

* patients that had undergone or will undergo a surgery under general anesthesia .

Exclusion Criteria:

* known history of syndromal craniofacial abnormalities (e.g. Down syndrome)
* previous craniofacial surgery
* excessive facial hair which significantly obscure facial landmarks
* cervical spine fractures
* tracheostomy tube
* patients who are unable to give consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Wojtczak, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period for this study is from 11-3-2010 to 10-1-2012 done in a medical clinic setting.
Pre-assignment Details: Enrollment goal for this study was met so the study was closed.
Groups:
- Difficult Intubation Patients: Obese and morbidly obese patients with a large neck circumference. This arm was patients who were difficult to intubate during previous anesthetics provided by the staff anesthesiologists.
  3D Laser Scanning of the Head, measurements and digital photos of the neck and ultrasound of the tongue were performed.
- Control: Obese and morbidly obese patients with a large neck circumference. The control group will consist of patients with easy laryngoscopy and intubation, recruited prospectively.
  3D Laser Scanning of the Head, measurements and digital photos of the neck and ultrasound of the tongue were performed.
Period: Overall Study
Arm/Group | Difficult Intubation Patients | Control
Started | 12 | 16
Completed | 12 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Males and Females 18 years and older
Groups:
- Total: Total of all reporting groups
Arm/Group | Difficult Intubation Patients | Control | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 16 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Hyomental Distance Ratio
Description: A curved low-frequency transducer and a Flex focul 400 ultrasound system were used to visualize the tongue and shadows of the hyoid bone and mandible. Midsagittal and coronal/transverse scans from the ultrasound were analyzed using ImageJ. The hyomental distances in the neutral and heal-extended positions were measured from the upper border of the hyoid bone to the lower border of the mentum. The ratio is defined as the ratio of the hyomental distance at the extreme of head extension to that in the neutral position.
Time Frame: end of study approximately one year
Population: only 6 patients in each group were analyzed because the remaining patients were not eligible for analysis based on a review of their electronic medical chart
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Difficult Intubation Patients | Control
Number analyzed (Participants) | 6 | 6
ratio | 1.14 (0.02) | 1.02 (0.01)

2. Secondary Outcome: Mean Tongue Volume
Description: The midsagittal scans were used to measure the cross-sectional area of the tongue. Transverse scans obtained in the midsection of the tongue (at the glossal end of the genioglossus muscle) provided a measure of the tongue width, which was measured between the most distant points on its upper surface. The tongue volume was derived from the multiplication of the midsagittal cross-sectional area by the tongue width.
Time Frame: end of study approximately one year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Difficult Intubation Patients | Control
Number analyzed (Participants) | 6 | 6
cubic centimeters | 137 (29) | 168 (34)

ADVERSE EVENTS:
Arm/Group | Difficult Intubation Patients | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 0/12 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes